CLINICAL TRIAL: NCT02708771
Title: Effect of W-3 Polyunsaturated Fatty Acids on Serum Albumin Concentration in Patients With Acute Heart Failure, Hypoalbuminemia, and High Inflammatory Activity
Acronym: PROTEICA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital San Juan de la Cruz (Other)
Responsible Party: Principal Investigator, Juan Luis Bonilla Palomas, Head of Cardiology, Hospital San Juan de la Cruz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSJC-CAR-01-2015
Record Dates: First submitted 2016-03-06; First posted 2016-03-15 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): 4 daily capsules of polyunsaturated fatty acids omega-3, during 4 weeks. Each capsule contains: 460 mg eicosapentaenoic acid ethyl ester and 380 mg docosahexaenoic acid ethyl ester.
  Interventions: Drug: Polyunsaturated fatty acids omega-3
- Control (Placebo Comparator): Capsules of similar appearance and flavor without active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Polyunsaturated fatty acids omega-3 — 4 daily capsules of polyunsaturated fatty acids omega-3, during 4 weeks. Each capsule contains: 460 mg eicosapentaenoic acid ethyl ester and 380 mg docosahexaenoic acid ethyl ester.
  Arms: Intervention
Drug: Placebo — 4 daily capsules of similar appearance and flavor without active ingredient
  Other Names: Control
  Arms: Control

SUMMARY:
Assess whether high doses of ?-3 fatty acids added to standard treatment of patients with acute hearta failure, hypoalbuminemia and high inflammatory activity, promotes an increase in serum albumin

DETAILED DESCRIPTION:
Assess whether high doses of ?-3 fatty acids added to standard treatment of patients with acute hearta failure, hypoalbuminemia and high inflammatory activity, promotes an increase in serum albumin

Assess the effect of high doses of ?-3 fatty acids added to standard treatment of patients with acute hearta failure, hypoalbuminemia and high inflammatory activity on:

* Inflammatory activity (C-reactive protein)
* The development of biomarkers (NTproBNP).
* The prognosis of patients evaluated by the combined event of death from any cause or readmission for heart failure within three months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or olders hospitalized for acute heart failure, chronic decompensated or new onset of any etiology, presenting hypoalbuminemia (serum albumin ?3,4 g / dl) and high inflammatory activity (CRP ?2,5 mg / dl).

Exclusion Criteria:

* Impending doom
* Participating in other clinical trials
* Treatment with ?-3 acids in the last month prior to admission
* Percutaneous or surgical treatment of the cause of heart failure during hospitalization.
* Pregnant women.
* Renal failure on dialysis.
* Chronic liver disease Child-Pugh B or C.
* Acute infectious process.
* Active malignant neoplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-03; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Serum albumin levels | Four weeks
  Serum albumin levels in the fourth week

SECONDARY OUTCOMES:
C-reactive protein levels | Four weeks
  C-reactive protein levels in the fourth week
NTproBNP levels | Four weeks
  NTproBNP levels in the fourth week
Combined event of death from any cause or readmission for heart failure | Three months
  Combined event of death from any cause or readmission for heart failure within three months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Juan de la Cruz, Úbeda, Jaen, Spain